CLINICAL TRIAL: NCT03474601
Title: Seoul National University Pituitary Disease Cohort Study
Acronym: SNU-PIT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jung Hee Kim, Principal Investigator, Seoul National University Hospital
Other Study IDs: 1503-040-654
Record Dates: First submitted 2018-03-10; First posted 2018-03-22 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2019-03

CONDITIONS: Pituitary Disease; Pituitary Incidentaloma; Acromegaly; Central Diabetes Insipidus; Pituitary Stalk Compression Hyperprolactinaemia; Cushing's Disease; Pituitary Tumor; Prolactinoma
Keywords: Pituitary Diseases; Pituitary incidentaloma; Central Diabetes Insipidus; Pituitary Neoplasms
MeSH Terms: conditions — Pituitary Diseases; Acromegaly; Diabetes Insipidus, Neurogenic; Pituitary ACTH Hypersecretion; Pituitary Neoplasms; Prolactinoma | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood Pituitary tumor tissue
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- Acromegaly: Patients diagnosed with acromegaly
  Interventions: Other: Dynamic hormone study and Magnetic resonance imaging
- Cushing's disease: Patients diagnosed with Cushing's disease
  Interventions: Other: Dynamic hormone study and Magnetic resonance imaging
- Hyperprolactinemia/prolactinomas: Patients diagnosed with hyperprolactinemia/prolactinoma
  Interventions: Other: Dynamic hormone study and Magnetic resonance imaging
- Pituitary stalk lesions: Patients diagnosed with pituitary stalk lesions
  Interventions: Other: Dynamic hormone study and Magnetic resonance imaging
- Nonfunctioning pituitary adenomas: Patients diagnosed with nonfunctioning pituitary adenomas
  Interventions: Other: Dynamic hormone study and Magnetic resonance imaging
- Central diabetes insipidus: Patients diagnosed with central diabetes insipidus
  Interventions: Other: Dynamic hormone study and Magnetic resonance imaging
- Craniopharyngioma: Patients diagnosed with craniopharyngiomas
  Interventions: Other: Dynamic hormone study and Magnetic resonance imaging
- Others: Patients diagnosed with other suprasellar/parasellar lesions
  Interventions: Other: Dynamic hormone study and Magnetic resonance imaging

INTERVENTIONS:
Other: Dynamic hormone study and Magnetic resonance imaging — 1. Medical history
  2. Imaging examination including brain magnetic resonance imaging
  3. Blood (Basal hormone study and follow-up study) and pituitary tumor tissue

SUMMARY:
The purpose of this study is to investigate the treatment and natural history of pituitary disease. We have a longstanding interest in pituitary disease including acromegaly, central diabetes insipidus, and nonfunctioning pituitary adenoma. We will continue to follow patients and recruit new patients for treatment and follow-up. Blood and pituitary tumor tissue (when available through clinical care) will be saved for future analyses related to pituitary disease.

DETAILED DESCRIPTION:
Subjects for this study will be recruited if they are:

1. Adults, male or female aged 18 years or older
2. Have been diagnosed with pituitary diseases

ELIGIBILITY:
Inclusion Criteria:

* Subjects for this study will be recruited if they are:

  1. Adults, male or female aged 18 years or older
  2. diagnosed with pituitary diseases such as acromegaly, Cushing's disease, hyperprolactinemia, nonfunctioning pituitary adenoma, pituitary stalk lesions, central diabetes insipidus, and craniopharyngiomas

Exclusion Criteria:

* Patients who do not agree with the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with pituitary disease at Seoul National University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2015-03-15 (Actual); Primary Completion 2025-02-14 (Estimated); Study Completion 2025-02-14 (Estimated)

PRIMARY OUTCOMES:
Treatment outcome of pituitary diseases | Up to 10 years
  Remission rate

SECONDARY OUTCOMES:
Complications of pituitary disease | Up to 10 years
  Visual field defect or hypopituitarism, hormone hyperfunction-related complications

CONTACTS AND LOCATIONS:
Overall Officials: Jung Hee Kim, M.D, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No